CLINICAL TRIAL: NCT04468854
Title: Influence of the Dietary Supplement Luteolin on Memory in Healthy Subjects
Brief Title: Influence of Luteolin on Memory in Healthy Subjects
Acronym: LuMus-Basel 20
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Corona-Virus Lockdown (16th March in Switzerland)
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Prof. Dominique de Quervain, MD, Director Divicion of Cognitive Neuroscience, University of Basel
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019-01356
Record Dates: First submitted 2020-06-26; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Memory
MeSH Terms: interventions — Luteolin

STUDY DESIGN:
Intervention Model Description: * randomized
  * double-blind
  * placebo-controlled
  * cross-over
  * counter-balanced
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): In the experimental phase we will administer 500 mg Luteolin (2x250 mg capsules) per day formulated for oral administration for 7.5 days (first intake: visit 1/3 in the morning; last intake: visit 2/4 in the morning). The last intake on visits 2 resp. 4 is important as the participants then have to recall the learned material from visits 1 resp. 3 during a steady-state status of Luteolin.
  Interventions: Dietary Supplement: Luteolin
- Control Intervention (Placebo Comparator): Control intervention consists of identical looking placebo capsules containing mannitol formulated for oral administration to be taken twice daily (e.g. every morning and evening) for 7.5 days (first intake: visit 1/3 in the morning; last intake: visit 2/4 in the morning) with water.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Luteolin — Luteolin extracted from Chrysanthemum Ramat 98% HPLC by Scyherb® food grade certified according to Safe Quality Foods (SQF) - Level 3 Comprehensive Food Safety and Quality Management System Certification by the Safe Quality Food Institute (SQFI).
  Arms: Experimental intervention
Other: Placebo — mannitol formulated for oral administration (capsules)
  Arms: Control Intervention

SUMMARY:
Proof of concept study on physiological processes (forgetting and memory functions, attention, working memory) in participants after multiple administration of the dietary supplement Luteolin.

DETAILED DESCRIPTION:
In the experimental phase the investigator will administer 500 mg Luteolin (2x250 mg capsules) per day formulated for oral administration for 7.5 days (first intake: visit 1/3 in the morning; last intake: visit 2/4 in the morning). The last intake on visits 2 resp. 4 is important as the participants then have to recall the learned material from visits 1 resp. 3 during a steady-state status of Luteolin.

Subjects will be randomly allocated to treatment groups (starting with investigational product or placebo).

Identity of Investigational Product: Luteolin extracted from Chrysanthemum Ramat 98% HPLC by Scyherb® food grade certified according to Safe Quality Foods (SQF) - Level 3 Comprehensive Food Safety and Quality Management System Certification by the Safe Quality Food Institute (SQFI).

Control intervention consists of identical looking placebo capsules containing mannitol formulated for oral administration to be taken twice daily (e.g. every morning and evening) for 7.5 days (first intake: visit 1/3 in the morning; last intake: visit 2/4 in the morning) with water.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* healthy
* normotensive (BP between 90/60mmHg and 140/90mmHg)
* BMI <30 kg/m2
* aged between 18 and 40 years
* native or fluent German-speaking
* able and willing to give written informed consent as documented by signature and comply with the requirements of the study protocol

Exclusion Criteria:

* Bodyweight <50 kg
* acute or chronic psychiatric disorder (e.g. major depression, psychoses, somatoform disorder, suicidal tendency)
* concomitant acute or chronic disease state (e.g. renal failure, hepatic dysfunction, cardiovascular disease, acute infections etc.)
* women who are pregnant or breast feeding
* intention to become pregnant during the course of the study
* known or suspected non-compliance, drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders
* participation in another study with investigational drug within the 30 days preceding and during the present study
* enrolment of the investigator, his/her family members, employees and other dependent persons
* participation in one of our previous studies using the same memory tests in the past 2 years
* Psychoactive drugs and alcoholic beverages 3 days (psychoactive drugs) resp. 12 hours (alcohol) before test visits 1-4.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Visual Memory Test | after 3 minutes, short delay (20 minutes), long delay (7 days): to assess differences between these time points
  Performance in a visual memory test (Rey-Osterrieth complex figure test (Rey 1941) and (Osterrieth 1944)). As parallel version the modified complex Taylor figure test (Hubley 2002).
  Participants will have to copy the complex figure of Rey Osterrieth. After 3 and 20 minutes delay the subject will be asked to draw the figure from memory. 7 days after learning there will be a delayed recall.
  Performance is calculated by scoring for accuracy and relative position of the 18 units in the whole of the design. Maximal score is 36 points.
Verbal Memory Task | immediate recall, short delay (15 minutes), long delay (7 days): to assess differences between these time points
  Verbal memory task (de Quervain, Roozendaal et al. 2000). A parallel version will be used for the second study phase.
  Subjects will view series of 60 unrelated German nouns each presented for 4 s on a computer screen with the explicit instruction to learn them for immediate and delayed recall. For the free-recall test, subjects will be asked to write down all the words they remember. The number of correctly recalled words (hits) will be the relevant output. Delayed recall of all 60 words will be tested about 15 min (short delay) and 7 days (long delay, after treatment phase) after presentation.

SECONDARY OUTCOMES:
Digit Span Task | after each treatment phase (duration one week) on vists 2 and 4
  Performance in a Working memory test assessed by the digit span task, a subtest of the WIE (von Aster 2006). A parallel version will be used for each visit. Each correct reproduction of a sequence of numbers is scored with one point.
Mode state (MDBF) | after each treatment phase (duration one week) on vists 2 and 4
  Mood state will be assessed for the past treatment phases of one week (visit 2 and 4) with the self-rating instrument MDBF (Steyer 1997) consisting of 12 items to be rated in a 5 scale mode. The total score is calculated by summing the answers in each of the 3 dimensions good/bad mood, alertness/sleepiness, rest /restlessness with 4 items in each dimension. We will use Version A and Version B.
Depressive symptoms | after each treatment phase (duration one week) on vists 2 and 4
  Depressive symptoms will be assessed with the self-rating questionnaire MADRS-S (Schmidtke 1988) for the past week (treatment phases). This scale consists of 9 items assessing participants' mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life. Each item is scored between 0 and 3. The total score is calculated by summing the answers of the nine items, ranging between 0 and 27 (higher scores indicate increased impairment).
Anxiety | after each treatment phase (duration one week) on vists 2 and 4
  Anxiety will be measured for the past treatment phases with the self-rating instrument STAI-G form X1 (state) (Laux 1981).This instrument consists of 20 items scored between 1-4. The total score is calculated by summing the answers, ranging between 20 and 80.
Visual Analog Scales Subjective Memory Function | after each treatment phase (duration one week) on vists 2 and 4
  Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm) between the two end-points: better memory function respectively than normal or worse. The score ranges between -5 and + 5.
Visual Analog Scales Quality of Sleep | after each treatment phase (duration one week) on vists 2 and 4
  Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm) between the two end-points: better sleep quality respectively than normal or worse. The score ranges between -5 and + 5.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, MD, Principal Investigator — University of Basel
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Canton of Basel-City, Switzerland